CLINICAL TRIAL: NCT02827136
Title: Ajou University School of Medicine
Brief Title: Effect of Lidocaine Patch for Shoulder Pain in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-16-076
Record Dates: First submitted 2016-07-04; First posted 2016-07-11 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases | interventions — hypafix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patch group (Experimental): Lidocaine patch and Hypafix
  Interventions: Drug: Lidocaine patch and hypafix
- Control group (Placebo Comparator): Just Hypafix
  Interventions: Drug: hypafix

INTERVENTIONS:
Drug: Lidocaine patch and hypafix — Appliance of Lidocaine patch and hypafix on both shoulder tip after anesthetic induction
  Arms: Patch group
Drug: hypafix — Appliance of hypafix on both shoulder tip after anesthetic induction
  Arms: Control group

SUMMARY:
The primary purpose of this study is to investigate the effect of lidocaine patch on the shoulder pain score after end of surgery.

The secondary purpose of this study is to investigate the effect of lidocaine patch on the total number of analgesic request on ward.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* Infection, trauma, or bleeding on shoulder
* Allergy to lidocaine
* Chronic pain
* Renal dysfunction
* Liver dysfunction
* Seizure
* History of shoulder surgery

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Shoulder pain score | Change from baseline shoulder pain score up to 24 hr after end of surgery

SECONDARY OUTCOMES:
Total number of analgesics request on ward | Up to postoperative day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, Seoum, South Korea